CLINICAL TRIAL: NCT06743984
Title: Shade Matching of Polychromatic Versus Monochromatic Composite Layering Techniques in Fractured Class IV Maxillary Central Incisors: a Randomized Clinical Trial
Brief Title: Evaluate the Shade Matching of Polychromatic Versus Monochromatic Composite Layering Techniques in Fractured Class IV Maxillary Central Incisors Using Universal , Layering & One Shade Composite In-vivo on Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Amira Mohammad Samy, Ass. Professor, Badr University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUC-IACUC-241117-117
Record Dates: First submitted 2024-12-02; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Class IV Dental Caries
Keywords: Universal resin composite; Monoshade resin composite; Polychromatic composite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single shade resin composite technique (Active Comparator): Nanohybrid single shade resin composite
  Interventions: Other: Polychromatic resin composite; Other: Monochromatic resin composite

INTERVENTIONS:
Other: Polychromatic resin composite — Polychromatic layering resin composite (enamel and dentin shades).
Other: Monochromatic resin composite — Monochromatic resin composite (opaquer and dentin shades)

SUMMARY:
The goal of this clinical trial is to evaluate shade matching ability of different techniques of application and different materials of resin composite restorations in class IV carious lesions

DETAILED DESCRIPTION:
Shade matching cabability of different resin composite materials and different techniques for restoration application, layering versus conventional incremental

ELIGIBILITY:
Inclusion Criteria:

1- Fractured class IV upper central incisors.

Exclusion Criteria:

1- cracked teeth

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
shade matching evaluation | 1 months
  evaluation of color change will be done using easy shade device & digital camera.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED A ABDELAZIZ, ASS. PROFESSOR, Study Director — BADR UNIVERSITY IN CAIRO
Locations (1):
- Badr University in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No